CLINICAL TRIAL: NCT07033897
Title: Adapting, Implementing and Evaluating the Effectiveness of the Home Hazard Removal Program for People With Disabilities
Brief Title: Adapting, Implementing and Evaluating the Effectiveness of HARP for People With Disabilities
Acronym: HARP3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202506116; MOHHU0088-24 (Other Grant/Funding Number: Department of Housing and Urban Development)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Disabilities Physical; Falls; Fall Prevention; Adults
Keywords: Fall prevention; Falls; People with disabilities; Adults; Home Hazard Removal Program; Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted HARP Intervention (Experimental): Participants in this group receive the adapted HARP intervention.
  Interventions: Behavioral: Adapted HARP
- Waitlist Control (No Intervention): Participants in this group receive virtual social visits. They will be offered the adapted HARP intervention after the 12-month follow-up visit is completed.

INTERVENTIONS:
Behavioral: Adapted HARP — The adapted HARP intervention includes two to three in-home visits conducted by an OT practitioner over approximately 5 weeks in the homes of PwD. At the end of the first home visit, solutions to remove the identified fall hazards will be determined collaboratively with the participant, using motivational interviewing to establish hazards and shared-decision making and tailoring to help the participant brainstorm solutions to remove the hazards. Participants will then receive one to two additional visits from the OT, and a contractor if needed, to implement solutions using a self-management approach, identifying any additional hazards and subsequent modifications if necessary. All adaptive equipment and modifications will be provided at no cost to the participant. Booster visit(s) will be completed 3-6 months after the initial treatment sessions to ensure the home modifications are still appropriate, troubleshoot any equipment issues and review the self-management process.
  Arms: Adapted HARP Intervention

SUMMARY:
The Home Hazard Removal Program (HARP) is an effective fall prevention intervention program which targets home hazard identification/removal. In this study the investigators will examine the effectiveness and implementation potential of HARP, adapted for PwD. Investigators will conduct a pilot randomized control trial (RCT) to test the implementation, cost, and preliminary efficacy of an adapted version of HARP for community-dwelling PwD. The single-blinded feasibility RCT will randomize 40 participants to treatment (adapted HARP) and 40 to a waitlist control group. Data on specific types of fall hazards and resulting home modifications as well as falls and fall-related injuries (collected monthly over 12 months) and fear of falling (collected at baseline and 12 months) will inform the preliminary efficacy of adapted HARP among PwD. To ensure usefulness, relevance, and broad dissemination of findings, the investigators will adopt a "designing for implementation and dissemination" approach. The RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework will guide intervention adaptation, trial design, and future implementation. The Practical Robust Implementation and Sustainability Model (PRISM) guides study development by identifying multi-level contextual factors hypothesized to affect the RE-AIM outcomes.

DETAILED DESCRIPTION:
The Home Hazard Removal Program (HARP) is an effective fall prevention intervention program which targets home hazard identification/removal, previously demonstrating a 38% reduction in falls among older adults with high fall risk. In this study investigators will examine the effectiveness and implementation potential of HARP, adapted for people with disabilities (PwD). The investigators will use a hybrid approach including a pilot RCT and a mixed methods study (semi-structured interviews and focus group) to adapt and examine the implementation and preliminary efficacy of HARP.

The investigators will conduct a Phase IIb pilot RCT study to test the feasibility and preliminary efficacy of an adapted version of HARP in community-dwelling PwD. The single-blinded RCT will randomize 40 participants to adapted HARP and 40 to waitlist control. Data on specific types of fall hazards and resulting home modifications as well as falls and fall-related injuries (collected monthly over 12 months) and fear of falling (collected at baseline and 12 months) will inform the preliminary efficacy of adapted HARP among PwD.

To ensure usefulness, relevance, and broad dissemination of findings, the investigators will adopt a "designing for implementation and dissemination" approach. The RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework, which guides planning and outcome evaluation of programming, will guide intervention adaptation, trial design, and future implementation. The Practical Robust Implementation and Sustainability Model (PRISM) has guided study development by identifying multi-level contextual factors hypothesized to affect the RE-AIM outcomes. Mixed methods using both quantitative and qualitive data (i.e., semi-structured interviews with 10 participants and a focus group with stakeholders [e.g., St. Louis Area Agency on Aging case managers, referral and evaluation specialists) will incorporate metrics from PRISM and RE-AIM, such as enrollment metrics, fidelity of implementation, number and specific location of fall hazards in the home, number, type and cost of home modifications, long-term adherence to home modifications and reduction in home hazards, qualitative perspectives on strengths and barriers, and willingness to adopt similar programming. Data will be used to identify the specific location of fall hazards, places where falls tend to occur in the home, and strategies to remediate these hazards.

ELIGIBILITY:
Inclusion Criteria:

* age 45-64 years
* self-report of difficulty with ≥2 daily activities
* have had a physical disability for ≥5 years (e.g., spinal cord injury, cerebral palsy, post-polio syndrome, stroke, amputation)
* live in the City of St. Louis
* had a fall in the past year, or are worried about falling, or feel unsteady when standing or walking

Exclusion Criteria:

• individuals who are institutionalized

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-03-14 (Estimated); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Falls | 12 months
  Reduction in fall rates

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Stark, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Final de-identified data will be preserved and shared with the public via WashU Research Data, an institutional repository managed by the Washington University in St. Louis Libraries. Datasets submitted to the data repository undergo curation prior to publication to ensure that the data are functioning, in the appropriate format, and well documented to facilitate long-term FAIRness (findable, accessible, interoperable and reusable). Submissions receive digital object identifiers minted with DataCite, and the library will retain the deposits for a minimum of 10 years.
Time Frame: Data will be available after the curation period for a minimum of 10 years
Access Criteria: De-identified data will be made available to the public